CLINICAL TRIAL: NCT04260516
Title: The Effect of N-acetylcysteine on Oxidative Stress Status and Iron Overload in Thalassemia Major
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Heba Mostafa Ahmed, Assistant Professor, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FM-BSU REC
Record Dates: First submitted 2020-02-04; First posted 2020-02-07 (Actual); Last update posted 2020-02-07 (Actual); Status verified 2020-02

CONDITIONS: Thalassemia Major
MeSH Terms: conditions — beta-Thalassemia | interventions — Acetylcysteine

STUDY DESIGN:
Intervention Model Description: Two groups are followed up for study parameters for 3 months one group is the intervention group and the other is the control group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- N-acetylcysteine group (Active Comparator): Patients received oral n-acetylcysteine syrup on dose of 10 mg/kg/day as single dose for 3 months
  Interventions: Drug: N-acetyl cysteine
- Non n-acetylcysteine group (No Intervention): Thalassemia major patients on regular chelation therapy who didn't receive n-acetylcysteine and served as controls

INTERVENTIONS:
Drug: N-acetyl cysteine — Mucolytic and antioxidant drug
  Arms: N-acetylcysteine group

SUMMARY:
The effect of N-acetylcysteine as antioxidant and its effect on pretransfusion hemoglobin and iron overload in patients with thalassemia were compared to patients who didn't receive n-acetylcysteine after 3 months of study duration

DETAILED DESCRIPTION:
N-acetylcysteine( NAC) is a widely used mucolytic drug and several studies had reported its efficacy as anti oxidant. Patients with thalassemia major are at great risk for oxidative stress due to excess of b-globin chains and iron overload. In this study the investigators compared the effect of NAC on oxidative status , pretransfusion hemoglobin levels and iron overload in thalassemia patients before and after treatment with NAC for 3 months and with that of patients who served as controls.

ELIGIBILITY:
Inclusion Criteria:

* Thalassemia major children on regular blood transfusion and iron chelation therapy

Exclusion Criteria:

* Renal or hepatic impairments
* Complicated thalassemia major
* Non adherence to therapy or follow up visits
* Change in the iron chelation dose within 3 months before enrollment or during study period

Ages: 3 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2019-06-03 (Actual); Primary Completion 2019-12-03 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Oxidative stress index (pg/mmol) | 3 months
  Oxidative stress index is calculated as the ratio of total oxidative status (pg/dl) to total anti oxidative capacity (mmol/dl)
Serum ferritin level ( mg/dl) | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Heba M Ahmed, Principal Investigator — Beni-Suef University
Locations (1):
- Heba Mostafa Ahmed, Banī Suwayf, Beni Suweif Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ozdemir ZC, Koc A, Aycicek A, Kocyigit A. N-Acetylcysteine supplementation reduces oxidative stress and DNA damage in children with beta-thalassemia. Hemoglobin. 2014;38(5):359-64. doi: 10.3109/03630269.2014.951890. Epub 2014 Sep 15. PMID 25222041